CLINICAL TRIAL: NCT04996706
Title: The Lymphoma Epidemiology of Outcomes (LEO) Cohort Study Protocol
Brief Title: Evaluation of Lymphoma Prognosis and Survivorship in Recently Diagnosed Patients, LEO Study
Acronym: LEO
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Emory University (Other); University of Iowa (Other); M.D. Anderson Cancer Center (Other); Washington University School of Medicine (Other); University of Rochester (Other); Weill Medical College of Cornell University (Other); University of Miami (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-001804; U01CA195568-06A1 (NIH); NCI-2022-02481 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphatic Diseases; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphatic Diseases; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood Collection
  2. DNA - Blood
  3. Tumor DNA and RNA Extraction
  4. Formalin Fixed Paraffin Embedded Tissue (FFPE) H&E Slide
  5. Tissue Microarrays (TMA)
  6. Clinical Residual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this infrastructure protocol is to build and maintain a large and diverse observational cohort study to support broad and cutting-edge research focused on NHL prognosis and survivorship. The LEO cohort will promote identification of clinical (including co-morbid diseases), epidemiologic (including lifestyle and other exposures), host genetic, tumor, and treatment factors that impact multiple outcomes (including event-free, overall and lymphoma-specific survival; new onset comorbidities; and patient-reported outcomes). This resource also will allow examination of the interaction among these factors in order to better understand the clinical and molecular epidemiology of outcomes in NHL. Ultimately, this approach will drive discovery and validation of treatment endpoints, improve prognostication, and identify novel approaches to improve short and long-term outcomes for NHL patients.

DETAILED DESCRIPTION:
1. To extend recruitment at all 8 LEO centers as part of LEO2.0 using a single IRB, with a goal of recruiting an additional 8,000 newly diagnosed NHL patients (with funding from the NIH renewal grant to enroll 3,400) focused on Hispanic (N=900), African Americans (N=580), and Asian (N=200) participants (doubling the current sample size for these groups; adolescent and young adult patients age 18-39 years (N=870; 87% increase); and non-metro and rural patients of all ages and race/ethnicities (N=1,208, 72% increase) for a total cohort of over 21,000 patients;
2. To review pathology at diagnosis and relapse of all LEO cases and maintain a central tumor bank for selected NHL subtypes that includes an H&E slide, formalin-fixed, paraffin-embedded (FFPE) tissue samples in a tissue microarray (TMA), and extracted tumor DNA and RNA;
3. To collect a peripheral blood sample and maintain a central biorepository of DNA, serum, plasma, and buffy coat;
4. To continue to prospectively follow all participants in the LEO cohort to ascertain disease progression/relapse, retreatment, transformation, second cancers, survival (including cause of death), updated exposures, patient-reported outcomes (PROs), and other long-term health outcomes;
5. To annotate and harmonize all cases with clinical, epidemiologic, pathology and treatment data, including development of new informatics enhancements to capture clinical data from electronic health records (EHRs), digital pathology, and radiology images, geocoded data from residence at diagnosis with linkage to public databases to enhance data on environmental exposures and socioeconomic factors; and
6. Facilitate research projects that use this infrastructure, promote interactions with NCI-supported clinical trials networks, patient advocacy groups, and other collaborators, and to make the LEO resource accessible to patients and providers with publicly available risk calculators based on LEO data.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-Hodgkin Lymphoma (NHL), within 183 days of enrollment
* Patients may have been treated as long as initial NHL diagnosis is within 6 months of enrollment
* 18 years of age or older

Exclusion Criteria:

- Lymphoma diagnosis greater than 184 days from date of consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed non-Hodgkin Lymphoma willing to provide a research blood sample, return enrollment and follow-up questionnaires, and allow access to medical records.
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Time Frame: Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of death

SECONDARY OUTCOMES:
Event Free Survival (EFS) | Time Frame: Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of first defined event (disease progression, relapse or re-treatment for lymphoma, or death)
Lymphoma Specific Survival (LSS) | Time Frame: Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of death due to lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: James R Cerhan, MD,PhD, Principal Investigator — Mayo Clinic
Locations (10):
- United States (10):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami: Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data can be requested through the LEO Cohort website.
Supporting Information: Study Protocol, SAP
Time Frame: Will become available upon publication
Access Criteria: Data sharing can occur only after going through group approvals.
URL: https://leocohort.org/

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials